CLINICAL TRIAL: NCT02487953
Title: Electronic Nicotine Delivery Systems (ENDS) as a Smoking Cessation Treatment
Brief Title: Electronic Nicotine Delivery Systems as a Smoking Cessation Treatment
Acronym: ENDS-P50
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study design changed significantly; was submitted as a different protocol.
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00063900; P50DA027840 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking; Smoking cessation; Nicotine patches; E-cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Cessation; Vaping | interventions — Tobacco Use Cessation Devices; Nicotine; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Nicotine ENDS + Nicotine Patch (Experimental): Participants will initially receive 1 week of 21 mg nicotine skin patches while continuing to smoke their usual cigarettes ad lib. Starting with week 2, they will receive nicotine-containing ENDS devices and will be instructed to substitute ENDS for as many cigarettes as possible in this week. The target quit-smoking date will occur at the beginning of week 3. Treatments will continue until week 8 post-quit, at which time participants will be instructed to reduce ENDS use over the next 4 weeks, at which time ENDS will no longer be dispensed. Subsequently, the nicotine patch dose will be gradually reduced according to standard weaning regimen from 21 mg/24 h to 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks. All nicotine-based treatments will end at week 16 after the quit date.
  Interventions: Drug: Nicotine patch; Other: ENDS
- Nicotine ENDS + Placebo Patch (Active Comparator): Participants will initially receive 1 week of placebo skin patches while continuing to smoke their usual cigarettes ad lib. Starting with week 2, they will receive nicotine-containing ENDS devices and will be instructed to substitute ENDS for as many cigarettes as possible in this week. The target quit-smoking date will occur at the beginning of week 3. Treatments will continue until week 8 post-quit, at which time participants will be instructed to reduce ENDS use over the next 4 weeks, at which time ENDS will no longer be dispensed. Subsequently, the placebo patch size will be gradually reduced to mirror standard weaning regimen from 21 mg/24 h to 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks. All nicotine-based treatments will end at week 16 after the quit date.
  Interventions: Other: ENDS; Other: Placebo patch
- Placebo ENDS + Nicotine Patch (Active Comparator): Participants will initially receive 1 week of 21 mg nicotine skin patches while continuing to smoke their usual cigarettes ad lib. Starting with week 2, they will receive placebo ENDS devices and will be instructed to substitute ENDS for as many cigarettes as possible in this week. The target quit-smoking date will occur at the beginning of week 3. Treatments will continue until week 8 post-quit, at which time participants will be instructed to reduce ENDS use over the next 4 weeks, at which time ENDS will no longer be dispensed. Subsequently, the nicotine patch dose will be gradually reduced according to standard weaning regimen from 21 mg/24 h to 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks. All nicotine-based treatments will end at week 16 after the quit date.
  Interventions: Drug: Nicotine patch; Other: Placebo ENDS

INTERVENTIONS:
Drug: Nicotine patch — 21 mg/24 h for 2 weeks before the quit date and 12 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks.
  Other Names: Nicoderm
  Arms: Nicotine ENDS + Nicotine Patch; Placebo ENDS + Nicotine Patch
Other: ENDS — As needed for 1 week before the quit date and 8 weeks after the quit date, then reduced use for 4 weeks.
  Other Names: e-cigarettes
  Arms: Nicotine ENDS + Nicotine Patch; Nicotine ENDS + Placebo Patch
Other: Placebo patch — 21 mg size for 2 weeks before the quit date and 12 weeks after the quit date, 14 mg size for 2 weeks, and 7 mg size for 2 weeks.
  Arms: Nicotine ENDS + Placebo Patch
Other: Placebo ENDS — As needed for 1 week before the quit date and 8 weeks after the quit date, then reduced use for 4 weeks.
  Arms: Placebo ENDS + Nicotine Patch

SUMMARY:
The purpose of this research study is to determine whether combining electronic nicotine delivery systems (ENDS) with nicotine patch treatment will augment abstinence rates compared to either treatment alone.

DETAILED DESCRIPTION:
Cigarette smokers, who are motivated to quit smoking but who rate the inhalation aspects of smoking as important will be randomized to three groups: Group 1. Nicotine ENDS + nicotine patch; Group 2: Nicotine ENDS + placebo patch; Group 3: Placebo ENDS + Nicotine patch. Participants will initially receive 1 week of 21 mg nicotine (or placebo) skin patches while continuing to smoke their usual cigarettes ad lib, in order to assess responsiveness to Nicotine Replacement Therapy (NRT). Starting with week 2, participants will receive nicotine-containing (or placebo) ENDS devices (menthol or non-menthol versions in accordance with their baseline preference). They will also be instructed to substitute ENDS for as many cigarettes as possible in this week. The target quit-smoking date will occur at the beginning of week 3. Treatments will continue until week 8 post-quit, at which time participants will be instructed to reduce ENDS use over the next 4 weeks, at which time ENDS will no longer be dispensed. Subsequently, the nicotine patch dose will be gradually reduced according to standard weaning regimen from 21 mg/24 h to 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks. All nicotine-based treatments will end at week 16 after the quit date.

ELIGIBILITY:
Inclusion Criteria:

* Have no known serious medical conditions;
* Smoke an average of at least 10 cigarettes per day;
* Have an expired air CO reading of at least 15 ppm;
* Able to read and understand English;
* Express a desire to quit smoking in the next thirty days;
* Higher than median rating of enjoyment of airway sensory effects of inhaling smoke on Cigarette Evaluation Questionnaire.

Exclusion Criteria:

* Hypertension;
* Hypotension;
* Coronary heart disease;
* Lifetime history of heart attack;
* Cardiac rhythm disorder (irregular heart rhythm);
* Chest pains (unless history, exam, and ECG clearly indicate a non-cardiac source);
* Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
* History of skin allergy;
* Active skin disorder (e.g., psoriasis) within the last five years;
* Liver or kidney disorder (except kidney stones, gallstones);
* Gastrointestinal problems or disease other than gastroesophageal reflux or heartburn;
* Ulcers;
* Lung disorder/disease (including but not limited to Chronic obstructive pulmonary disease (COPD), emphysema, and asthma);
* Brain abnormality (including but not limited to stroke, brain tumor, and seizure disorder);
* History of migraine headaches in the past 5 years;
* History of fainting;
* Problems giving blood samples;
* Difficulty passing urine;
* Diabetes treated with insulin; non-insulin treated diabetes (unless glucose is less than 180mg/dcl and HbA1c is less than 7%);
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition;
* Current psychiatric disease (with the exception of anxiety disorders, Obsessive Compulsive Disorder (OCD) and ADHD);
* Suicidal ideation (within the past 10 years) or lifetime occurrence of attempted suicide;
* Current depression;
* Bulimia or anorexia;
* Pregnant or nursing mothers;
* Use (within the past 30 days) of:

  * Illegal drugs (or if the urine drug screen is positive for tetrahydrocannabinol (THC), Cocaine, Amphetamine, Opiates, Methamphetamines, phencyclidine (PCP), Benzodiazepines, or Barbiturates),
  * Experimental (investigational) drugs;
  * Psychiatric medications including antidepressants, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
  * Smokeless tobacco (chewing tobacco, snuff), cigars, pipes, nicotine replacement therapy, e-cigarettes or other smoking cessation treatment;;
* Alcohol abuse;
* Significant adverse reaction to nicotine patches in the past;
* Current participation or recent participation (in the past 30 days) in another smoking study at our Center or another research facility;
* Current participation in another research study.

Potential subjects must agree to use acceptable contraception.

Potential subjects must agree to avoid the following:

* participation in any other nicotine-related modification strategy outside of this protocol;
* use of tobacco products other than cigarettes, including pipe tobacco, cigars, e-cigarettes, snuff, and chewing tobacco;
* use of experimental (investigational) drugs or devices;
* use of illegal drugs;
* use of opiate medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Continuous four-week abstinence from smoking during treatment | Weeks 4-8 post target Quit Day
  The primary outcome measure will be continuous four-week abstinence from smoking during weeks 4-8 post target Quit Day while treatment is ongoing. This will be determined by a composite of self-report of no smoking on daily diaries and expired air carbon monoxide (CO) <10 ppm (measured at Week 8). An intent-to-treat criterion will be used, whereby drop-outs are considered to be non-abstinent.

SECONDARY OUTCOMES:
Continuous four-week abstinence from smoking after withdrawal of ENDS | Weeks 9-12 post target Quit Day
  A secondary outcome measure will be continuous four-week abstinence from smoking during weeks 9-12 post target Quit Day while participants are decreasing their use of ENDS. This will be determined by a composite of self-report of no smoking on daily diaries and expired air carbon monoxide (CO) <10 ppm (measured at Week 12). An intent-to-treat criterion will be used, whereby drop-outs are considered to be non-abstinent.
Continuous four-week abstinence from smoking after withdrawal of nicotine patches | Weeks 13-16 post target Quit Day
  A secondary outcome measure will be continuous four-week abstinence from smoking during weeks 13-16 post target Quit Day while participants are using decreasing doses of nicotine patches. This will be determined by a composite of self-report of no smoking on daily diaries and expired air carbon monoxide (CO) <10 ppm (measured at Week 16). An intent-to-treat criterion will be used, whereby drop-outs are considered to be non-abstinent.
Seven-day point abstinence from smoking at 6 months post Quit Day | 6 months post Quit Day
  A secondary outcome measure will be seven-day abstinence from smoking at six months post target Quit Day. This will be determined by self-report of no smoking for the previous seven days when called for 6-month follow-up, verified by expired air carbon monoxide (CO) <10 ppm (measured at 6-month follow-up visit). An intent-to-treat criterion will be used, whereby drop-outs are considered to be non-abstinent.

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University; James M Davis, M.D., Principal Investigator — Duke University
Locations (1):
- Duke Center for Smoking Cessation, Durham, North Carolina, United States